CLINICAL TRIAL: NCT05011643
Title: The Effects of Statins on Muscle Damage Markers After Moderate-intensity Exercise
Brief Title: Exercise-induced Muscle Damage in Statin Users
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: CMO 2007-148
Record Dates: First submitted 2021-08-15; First posted 2021-08-18 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Cardiovascular Diseases; HMG COA Reductase Inhibitor Adverse Reaction; Muscle Damage
Keywords: Statin-associated muscle symptoms; Muscle damage markers; Moderate-intensity exercise; Coenzyme Q10
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples to analyze muscle damage markers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Symptomatic statin users: Statin users with self-reported muscle symptoms
  Interventions: Other: Moderate-intensity exercise
- Asymptomatic statin users: Statin users without muscle symptoms
  Interventions: Other: Moderate-intensity exercise
- Non-statin using controls: Participants not using statins
  Interventions: Other: Moderate-intensity exercise

INTERVENTIONS:
Other: Moderate-intensity exercise — Participants will walk either 30km, 40km or 50km for four consecutive days during the Nijmegen Four Days Marches. Measurements will be performed after the finish of the first, second and third walking day.

SUMMARY:
Rationale: Combining statin treatment and physical activity is very effective for the prevention of cardiovascular diseases. Statins are well-tolerated by most patients, but may cause statin-associated muscle symptoms (SAMS) and elevated markers of skeletal muscle damage in some patients.

Several studies have shown that statins augment increases in serum creatine kinase after eccentric or vigorous exercise. If statins also increase muscle damage markers after exercises of moderate intensity is unclear. Symptomatic statin users may be more susceptible to exercise-induced skeletal muscle injury, however, previous studies did not differentiate between symptomatic and asymptomatic statin users.

Objective: To compare the impact of moderate-intensity exercise on muscle damage markers between symptomatic and asymptomatic statin users, and non-statin using controls. A secondary objective is to examine the association between leukocytes coenzyme Q10 levels and exercise-induced muscle damage and muscle complaints.

DETAILED DESCRIPTION:
Combining statin treatment and physical activity is very effective for the prevention of cardiovascular diseases. Statins are well-tolerated by most patients, but may cause statin-associated muscle symptoms (SAMS) and elevated markers of skeletal muscle damage in some patients.

Several studies have shown that statins augment increases in serum creatine kinase after eccentric or vigorous exercise. However. if statins also increase muscle damage markers after exercises of moderate intensity is unclear. Impaired mitochondrial oxidative function might contribute to SAMS and exercise-induced muscle damage. Several studies showed that statins decrease serum coenzyme Q10 levels, an essential component of the mitochondrial transport chain, but effects on intramuscular coenzyme Q10 levels are inconsistent. The investigators have observed that mitochondrial dysfunction is more pronounced in statin users with SAMS compared to asymptomatic statin users. This suggests that symptomatic statin users may be more susceptible to exercise-induced skeletal muscle injury. However, previous studies examining creatine kinase response to exercise did not differentiate between symptomatic and asymptomatic statin users.

In this cross-sectional observational study the investigators will study the impact of moderate-intensity exercise on muscle damage markers between symptomatic and asymptomatic statin users, and non-statin using controls. A secondary objective is to examine the association between leukocytes coenzyme Q10 levels and exercise-induced muscle damage and muscle complaints.

The investigators hypothesize that statins will not increase muscle damage markers after moderate-intensity exercise and that higher CoQ10 levels are associated with less exercise-induced muscle damage and muscle complaints.

ELIGIBILITY:
Inclusion Criteria:

* Mentally able to give informed consent
* Statin groups: statin treatment for at least 3 months

Exclusion Criteria:

* Known hereditary muscle defect
* Known mitochondrial disease
* Diabetes Mellitus
* Hypo- or hyperthyroidism
* Other diseases known to cause muscle symptoms (e.g. m. Parkinson or rheumatic diseases)
* Coenzyme Q10 supplementation

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Symptomatic statin users (n=35), asymptomatic statin users (n=34) and non-statin using controls (n=31).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
Muscle damage markers | Baseline (before exercise) and after three days of moderate-intensity walking exercise (measured each day)
  Change in muscle damage markers (creatine kinase, myoglobin, lactate dehydrogenase, troponin I and BNP) from baseline to post-exercise

SECONDARY OUTCOMES:
Muscle pain scores | Baseline (before exercise) and after three days of moderate-intensity walking exercise (measured each day)
  Muscle pain scores measured with the Brief Pain Inventory questionnaire (10 point scale with 0 representing no pain and 10 the worst pain imaginable)
Muscle strength and fatigue | Baseline (before exercise) and after one day of moderate-intensity walking exercise
  M. Quadriceps muscle strength and fatigue measured using electrical stimulation
Coenzyme Q10 levels | At baseline
  Coenzyme Q10 levels measured in leukocytes

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physiology, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Allard NAE, Janssen L, Lagerwaard B, Nuijten MAH, Bongers CCWG, Rodenburg RJ, Thompson PD, Eijsvogels TMH, Assendelft WJJ, Schirris TJJ, Timmers S, Hopman MTE. Prolonged Moderate-Intensity Exercise Does Not Increase Muscle Injury Markers in Symptomatic or Asymptomatic Statin Users. J Am Coll Cardiol. 2023 Apr 11;81(14):1353-1364. doi: 10.1016/j.jacc.2023.01.043. PMID 37019582